CLINICAL TRIAL: NCT02424591
Title: A Prospective, Randomized, Single Blinded Comparison of Intraoperative Ketamine Infusion Versus Placebo in Patients Having Spinal Fusion
Brief Title: A Comparison of Intra-op Ketamine vs Placebo in Patients Having Spinal Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-00599
Record Dates: First submitted 2015-04-02; First posted 2015-04-23 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
Keywords: Anesthesia Recovery Period; Spinal Fusion
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): ketamine group will be infused after intubation and terminated at the start of skin closure
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): placebo group will have standard of care rather than ketamine infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — Infusion at a rate of 10 mcg/kg/min
  Other Names: Ketalar
  Arms: Ketamine
Other: Placebo — Placebo IV
  Arms: Placebo

SUMMARY:
Postoperative pain is severe after major spine surgery. Opioids such as morphine and hydromorphone are routinely used for postoperative pain control. These drugs have significant side effects, most importantly respiratory depression, nausea, constipation and tolerance. Moreover, many spine surgery patients have used opioid pain medication for back pain long term, leading to pre-surgical opioid tolerance and increased postoperative pain. This has led to a search for adjuvant medications to reduce the use of opioids and reduce opioid mediated side effects and tolerance.

Ketamine is an intravenous anesthetic with analgesic properties in subanesthetic doses. Ketamine is a noncompetitive antagonist of N-methyl-D-aspartate (NMDA) receptors. NMDA receptors are involved in central pain sensitization via wind-up phenomenon and altered pain memory, a process which can be blocked by ketamine. NMDA receptor antagonists may prevent the development of tolerance to opioids and hyperalgesia. Ketamine has been safely used to decrease pain in numerous studies. Ketamine can also act as an antidepressant with hours of administration.

Ketamine has rapid brain uptake and subsequent re-distribution with a distribution half-life of 10-15 minutes and an elimination half-life of 2 hours. Ketamine does not cause respiratory depression.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, placebo controlled single center trial. One hundred subjects (50 in each arm) will be enrolled. Subjects undergoing multilevel spinal fusion will be screened and have the study introduced and discussed with them during the preadmission visit. Subjects may also contact study personnel or be contacted by study personnel before admission. Upon admission on the day of surgery, patients will be re-screened, recruited, have informed consent obtained. After consent is achieved in the pre-admission clinic prior to surgery, patients will be asked to fill out Beck's depression inventory (BDI), post-operative quality of recovery score(QoR-15) form, visual analog scale (VAS) for pain and short form McGill pain questionnaire to establish baseline scores. These forms can be completed at pre-admission testing, at home or on the day of surgery. The three forms will be on postoperative days (POD) 1, 2 and 3; only the VAS will be given in the Post-Anesthesia Care Unit (PACU). Eligible subjects will be assigned to either the ketamine or placebo group based on a computer generated randomization (randomization.com). Baseline demographic data as well as medical history and medication list will be recorded.

Anesthetic management for this study will be exactly the same management that we are currently providing for patients undergoing multilevel spinal fusions. The only difference in care between the placebo group and the treatment group will be the addition of a low dose ketamine infusion in the treatment group. The placebo group will receive a fentanyl infusion at 1 mcg/kg/hr during the surgery and a morphine PCA for postoperative pain control. The placebo group will receive additional fentanyl as needed on the operating room and additional morphine as needed in the recovery room.

Anesthetic management for both groups will start with IV placement and routine (American Society of Anesthesiologists - ASA ) monitors. An arterial catheter may be placed at the discretion of the attending anesthesiologist. After preoxygenation, general anesthesia will be induced with Propofol 1 to 2 mg/kg, fentanyl 1 to 2 mcg/kg, and rocuronium .6 mg/kg. Maintenance of anesthesia will be a propofol infusion starting at 150 mcg/kg/min, fentanyl 1 mcg/kg/hr. Additionally, the ketamine group will receive a ketamine infusion at a rate of 10 mcg/kg/min starting after intubation and terminated at the start of skin closure. All patients will be treated with zofran and ofirmev during surgical closing. Pre-induction midazolam will be administered at the discretion of the anesthesiologist. No NSAIDS will be given because of bleeding risk. Sevoflurane may be used for brief periods at the beginning and end of the procedure to cover times when total intravenous anesthesia (TIVA) is not practical, i.e. when moving or positioning the patient. Additional fentanyl and rocuronium boluses can be given as needed. Administration of corticosteroids per surgeon's request will be recorded. Anesthetics will be titrated to maintain a Bispectral (BIS) index of 40 to 60. Patients will be awakened, extubated and transferred to the PACU after following simple commands. Morphine patient controlled anesthesia (PCA) at a setting of 1 mg dose with a 6 minutes lockout will be started immediately on arrival in PACU. While in the PACU, all subjects who do not have adequate pain control will receive rescue dose of morphine 2 mg. to 4 mg. as indicated by a numeric pain Rating Scale score > 3 or upon subjects' request. All narcotics and other pain medication given will be recorded. Postoperative nausea will be treated with droperidol .625 mg IV. If the patient's pain cannot be controlled with PCA morphine then a pain consult will be obtained. The pain service will be free to administer any medication deemed necessary to control the patient's pain.

PACU Monitoring: Once in the PACU, all patients will be monitored by PACU nurses per nursing protocol. The following questionnaires: 1) VAS for pain will be administered in the PACU. On postoperative day 1, 2 and 3 the McGill short form, VAS, Beck Depression Inventory (BDI) and QoR15 will be given.

The subjects who enroll in this study will be asked to fill out questionnaires at five different times. The questionnaires include The Beck depression inventory, McGill's short form pain questionnaire, Quality of Recovery - 15 form (QoR15) and the visual analog scale (VAS) for pain. The forms will be filled out at five separate times; preoperatively in pre-surgical testing or in the pre-surgical holding area of Tisch hospital, in the post anesthesia care unit of Tisch hospital after the surgery, on postoperative day #1, on postoperative day #2 and on postoperative day #3. In the PACU on the day of surgery, only the VAS will be given.

All subjects will be carefully monitored for safety and efficacy. While the ketamine or placebo is administered in the operating room, an anesthesiologist, Certified Registered Nurse Anesthetist (CRNA) or anesthesia resident will be present. In the PACU patients will have 1:1 or 1:2 nursing care. An anesthesiologist is immediately available in the PACU should a problem arise.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>/=18)
2. male or female
3. Undergoing surgery for multilevel (>2 level) spinal fusion from a posterior approach.
4. General anesthesia
5. English speakers such that they can complete the pain score and satisfaction questionnaires whose scores are a critical outcome variable.
6. If female, subject is non-lactating and is either: a. Post-menopausal or post hysterectomy; b. Of childbearing potential but is not pregnant at time of baseline as determined by pre-surgical pregnancy testing.
7. Subject is American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.

Exclusion Criteria:

1. Cognitively impaired (by history)
2. Subject with a history of psychosis
3. Subject known to have significant hepatic disease
4. Subject for whom opioids or ketamine are contraindicated
5. Patients with narrow angle glaucoma
6. Increased intracranial or intraocular pressure
7. If female, is either pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Ard, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Woolf CJ, Thompson SWN. The induction and maintenance of central sensitization is dependent on N-methyl-D-aspartic acid receptor activation; implications for the treatment of post-injury pain hypersensitivity states. Pain. 1991 Mar;44(3):293-299. doi: 10.1016/0304-3959(91)90100-C. PMID 1828878
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Perioperative ketamine for acute postoperative pain. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004603. doi: 10.1002/14651858.CD004603.pub2. PMID 16437490
- [Background] Machado-Vieira R, Salvadore G, Diazgranados N, Zarate CA Jr. Ketamine and the next generation of antidepressants with a rapid onset of action. Pharmacol Ther. 2009 Aug;123(2):143-50. doi: 10.1016/j.pharmthera.2009.02.010. Epub 2009 May 3. PMID 19397926
- [Background] Yamauchi M, Asano M, Watanabe M, Iwasaki S, Furuse S, Namiki A. Continuous low-dose ketamine improves the analgesic effects of fentanyl patient-controlled analgesia after cervical spine surgery. Anesth Analg. 2008 Sep;107(3):1041-4. doi: 10.1213/ane.0b013e31817f1e4a. PMID 18713926
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were approached either at pre-admission testing or at the peri-op area of the hospital. All patients were spoken to privately and given time to ask questions. After consent was signed, a copy was given to the subject and a copy put into the medical record.
Pre-assignment Details: One patient was excluded because his surgery was cancelled.
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 22 | 23
Completed | 20 | 20
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56 to 72] | 65 [53 to 72] | 65 [54 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 8 | 12 | 20
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Preoperative Opioid Use [Count of Participants; unit: Participants] | 9 | 8 | 17
Prior Back Surgery [Count of Participants; unit: Participants] | 11 | 13 | 24
Visual Analog Scale (VAS) Pain Score [Median (Inter-Quartile Range); unit: points] — The Visual Analog Scale is a way to measure pain, with zero being no pain at all and 10 being the most terrible pain.
  points | 7 [5 to 8] | 3.5 [2.8 to 7.0] | 6 [3 to 8]
American Society of Anesthesiologists Physical Status Score [Count of Participants; unit: Participants] — The American Society of Anesthesiologists Physical Status Score is assigned by the anesthesiologist at the time of providing care, based on the following definitions:
  ASA I - A normal healthy patient ASA II - A patient with mild systemic disease ASA III - A patient with severe systemic disease ASA IV - A patient with severe systemic disease that is a constant threat to life ASA V - A moribund patient who is not expected to survive without the operation ASA VI - A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    I | 0 | 1 | 1
    II | 10 | 8 | 18
    III | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Scores on Questionnaires
Description: Quality of Recovery 15 questions questionnaires that ask, on a scale of 0-10, with 0 always being bad and 10 always being best, how the patient is recovering. The total number is reviewed, so the highest total score possible is 150 and the lowest is 0.
Time Frame: Post-op Day 3
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
points | 95 [80 to 115.6] | 101 [86 to 109]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Score
Description: McGill Short Form measures pain in different ways. The first part of the form lists 15 adjectives for pain, for which the answers can be none (0), Mild (1), Moderate (2) and Severe (3). Descriptors 1-11 represent the sensory dimension of pain experience and 12-15 represent the affective dimension. A score of 0 is good, and a score of 45 indicates extreme pain. The lower the score the less pain a subject feels (better), as the scores go up, so do the pain levels (worse).
  PPI (Present Pain Intensity) asks patients to measure pain from 0 (no pain) to 5 (excruciating). Again, a lower score is ideal.
Time Frame: Post-op Day 3
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
points | 11 [4.5 to 18] | 10.5 [8 to 17]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Beck's Depression Inventory
Description: Beck's Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures attitudes and symptoms of depression. Each sentence has a rating from 0 to 3 and the sentences go from mild to fairly severe descriptions of moods. The numbers are tabulated, the lowest possible score is 0 and the highest is 63.
  A score of 1-10 indicates normal ups and downs. 11-16 indicates a mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; over 40, extreme depression
Time Frame: Post-op Day 3
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
points | 8 [5 to 16] | 9 [8 to 11]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data was reviewed for adverse events intraoperative through post-op day 3.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes